CLINICAL TRIAL: NCT02245893
Title: A Prospective Randomized Pilot Study to Compare Open Versus Percutaneous Syndesmosis Repair of Unstable Ankle Fractures
Acronym: ART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Sanders, Orthopedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103747
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Fracture Dislocation of Ankle Joint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screw (Active Comparator): In the SCREW Group (standard surgery technique), surgical treatment will be by closed reduction utilizing intraoperative fluoroscopy to visualize the reduction and percutaneous syndesmosis screw insertion. Intraoperative fluoroscopic stress and non-stress views will be obtained as per standard of care.
  'open reduction internal fixation (ORIF)
  Interventions: Procedure: open reduction internal fixation (ORIF)
- Anatomic repair technique (ART) (Active Comparator): In the ART group (study group) surgical treatment will be by open reduction and internal fixation. In order to stabilize the syndesmosis, direct visual anatomic alignment will be conducted and a syndesmotic screw inserted. In addition, fixation of the anterior ligament will be performed with use of a 2.7 to 4.0 mm suture anchor. Repair of the intact portion of the ligament will be made using a modified Mason -Allen repair. Intraoperative fluoroscopic stress and non-stress views will be obtained as per standard of care.
  'open reduction internal fixation (ORIF)
  Interventions: Procedure: open reduction internal fixation (ORIF)

INTERVENTIONS:
Procedure: open reduction internal fixation (ORIF) — The study design is a prospective, randomized pilot clinical trial of the treatment of unstable syndesmosis injuries sustained with Weber C type fractures. Comparison will be made between two syndesmosis stabilization methods: 1) Percutaneous (closed) reduction using syndesmosis fixation by SCREW 2) Open reduction (ORIF) with ART repair of the anterior ligament and stabilization of the syndesmosis by use of a syndesmosis screw.

SUMMARY:
This study evaluates fracture healing, anatomic reduction and return to functioning in patients with unstable Weber C type fractures of the ankle. Best outcomes are obtained when a good alignment of the ankle joint is maintained and natural function of the syndesmosis (space between the tibia and fibula bones) is restored. The syndesmosis and ankle joint is stabilized by a series of ligaments which are often damaged in Weber C type fractures. Current syndesmosis repair techniques traverse the tibia and fibula, but do not anatomically reconstruct the ligaments. The investigators will compare reconstruction of the unstable syndesmosis by open reduction and internal fixation using a syndesmosis screw coupled with anterior ligament (AiTFL) anatomic repair technique (ART) to percutaneous repair using a syndemosis screw only (SCREW). Radiographic, pain and functional outcome scores will be compared between the groups using validated outcome measures.

DETAILED DESCRIPTION:
High ankle fractures involve fracture of the fibula above the level of the syndesmosis (space between the tibia and fibula bones) that result from indirect mechanisms (e.g. pronation-external rotation (twisting) injuries. The method of injury is assumed to disrupt one or more of the syndesmotic ligaments, leading to instability of the ankle mortise . High ankle fractures comprise a significant proportion of ankle injuries (16 to 45 % of all ankle fractures patterns) . It is generally agreed that operative intervention of ankle injuries is indicated in cases of instability . However, recent advances in the understanding of the biomechanics of the ankle have given rise to particular areas of clinical uncertainty, including the treatment of unstable syndesmotic injuries and reliability of strictly radiographic assessment of ankle fractures .

The goal of operative treatment is to anatomically reduce the ankle mortise to permit syndesmosis ligament healing and restoration of the normal tibiofibular joint dynamics. Even 1 mm of displacement or lateral shift of the talus will affect ankle joint loading and lead to dysfunction and potentially degenerative joint changes. Accurate reduction of the syndesmosis and maintenance of this reduced position until the ligaments heal is crucial to ensure good outcome and to avoid long term arthritic changes in the tibiofibular joint .

If the ankle joint is unstable (too much sideways movement), the syndesmosis space between the two bones in the ankle (tibia and fibula) needs to be stabilized. One method to treat unstable syndesmosis injuries is making an incision to expose the ankle to provide direct visualization of fracture for anatomic reduction (alignment) and insertion of one or two syndesmosis screws to maintain the relationship of the fibula to the tibia. This is referred to as open reduction and internal fixation (ORIF).

Another method of repair is by closed reduction of the ankle joint and the use of one or two percutaneous syndesmosis screws only. That is, syndesmosis stabilization can be done percutaneously using intraoperative fluoroscopy to visualize the repair . Literature and standard practice support both of these methods.

The syndesmosis joint complex is composed of the anterior inferior tibiofibular ligament (AiTFL), the posterior inferior tibiofibular ligament (PiTFL) and the interosseous membrane (IOM). This complex is believed to permit ankle mortise stability and flexibility due to the elasticity of the ligaments, which allows the intermalleolar distance to change and facilitates tibial and fibular rotation. It also maintains the axis of balanced loading of the foot through the fibula. Adequate stability and anatomic restoration of the syndesmosis joint complex is vital to restoring normal tibiotalar contact forces in order to lessen the risk of posttraumatic arthritis.

Clinical studies have shown that anatomic reduction of the PiTFL provides a more accurate reduction of the ankle mortise than percutaneous reduction while ORIF fixation of the PiTFL has been shown on both biomechanical and clinical studies to provide greater stability than with syndesmotic screws alone .

However, due to the mechanism if injury, the AiTFL is the initial and may be the only lateral ligamentous stabilize structure compromised in syndesmotic injury. Kinematically, this ligament provides roughly half of the strength of the syndesmosis and acts as a vital primary restraint to excessive fibular displacement. The remainder of the stability is believed to come from bony restraints such as the posterior malleolus and the PiTFL . As such, direct reconstruction of the AiTFL component of the syndesmosis joint may accurately restore syndesmotic stability. Current syndesmosis repair techniques traverse the tibia and fibula (trans syndesmotic repair), but do not anatomically reconstruct the AiTFL.

Although it is known that an accurate reduction of the syndesmosis is essential to a good outcome, current treatments may have malreduction rates greater than 40% . In light of the existing models of syndesmosis injury, and the investigators' understanding of the importance of syndesmosis reduction, it may be that restoration of the AiTFL may potentially unlock a higher rate of anatomic reductions and positive outcomes.

Cadaveric and clinical studies have demonstrated that a flexible trans-osseous fixation technique may be viable and may improve ligamentous healing . However, current flexible techniques may not provide adequate stability and may not reduce the rate of malreduction compared to screw fixation.

The investigators recently conducted biomechanical studies in our lab using cadaveric ankles. The investigators compared whether a technique of syndesmosis repair concentrating on restoration of the AiTFL ligament (Anatomic repair technique or ART) provides a more anatomic reconstruction of the syndesmosis joint than rigid screw or posterior malleolus fixation.

The investigators' findings have demonstrated that our anatomic repair technique (ART) offers a repair which is sufficiently stable compared to screw fixation, with a lower incidence of malreduction as visualized on CT scan.

The investigator research suggests that ORIF repair of the AiTFL in addition to the stability provided by syndesmotic screw repair enhances syndesmosis stability substantially, as the AiTFL is a primary stabilizer to external rotation forces. In other words, fixing the anterior ligament may provide a better outcome and faster return to functioning.

Further in vivo testing is required to evaluate ART for repair of unstable syndesmosis injuries.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years old or greater with a pre-operative diagnosis of a Weber C ankle fracture (supination-external rotation, pronation-external rotation, pronation-abduction patterns).
2. The subject demonstrates lateral subluxation of the talus on x-ray or stress views (unstability).
3. The lateral malleolus fracture if present begins at least 1.0 cm proximal to the syndesmosis.
4. The subject has no history of previous ankle injury.
5. The subject does not have an ipsilateral lower extremity injury that would impede results.
6. The subject has no neuromuscular or neurosensory deficiency that would limit the ability to assess the operative procedure.

   -

Exclusion Criteria:

1. The subject has a lateral malleolus fracture that begins less than 1.0 cm proximal to the syndesmosis.
2. The subject has an open ankle fracture with a lateral wound. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
CT scan | 3 month
  assessment of ankle alignment

SECONDARY OUTCOMES:
Foot and Ankle Outcome Score (FAO), | 6 weeks, 3 , 6 , 12 months
  Functional outcome assessment
AOFAS Hindfoot Score | 6 weeks, 3 , 6 , 12 months
  Functional outcome assessment
Maryland Foot Score | 6 weeks, 3 , 6 , 12 months
  Functional outcome assessment
Radiographic healing | 6 weeks, 3 , 6 , 12 months
  xray
Complication- Infection | 6 weeks, 3 , 6 , 12 months
  clinical and xray review of fracture documented
Complication-Implant Failure | 6 weeks, 3 , 6 , 12 months
  clinical and xray review of fracture documented

CONTACTS AND LOCATIONS:
Overall Officials: David Sanders, Principal Investigator — Western Univeristy/Lawson Health ResearcH Institute
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris IA, Jones HP. The fate of the syndesmosis in type C ankle fractures: a cadaveric study. Injury. 1997 May;28(4):275-7. doi: 10.1016/s0020-1383(97)00010-7. PMID 9282181
- [Background] Leeds HC, Ehrlich MG. Instability of the distal tibiofibular syndesmosis after bimalleolar and trimalleolar ankle fractures. J Bone Joint Surg Am. 1984 Apr;66(4):490-503. PMID 6423645
- [Background] Ebraheim NA, Mekhail AO, Gargasz SS. Ankle fractures involving the fibula proximal to the distal tibiofibular syndesmosis. Foot Ankle Int. 1997 Aug;18(8):513-21. doi: 10.1177/107110079701800811. PMID 9278748
- [Background] Boden SD, Labropoulos PA, McCowin P, Lestini WF, Hurwitz SR. Mechanical considerations for the syndesmosis screw. A cadaver study. J Bone Joint Surg Am. 1989 Dec;71(10):1548-55. PMID 2512295
- [Background] Michelson JD. Fractures about the ankle. J Bone Joint Surg Am. 1995 Jan;77(1):142-52. doi: 10.2106/00004623-199501000-00020. No abstract available. PMID 7822349
- [Background] Solari J, Benjamin J, Wilson J, Lee R, Pitt M. Ankle mortise stability in Weber C fractures: indications for syndesmotic fixation. J Orthop Trauma. 1991;5(2):190-5. doi: 10.1097/00005131-199105020-00012. PMID 1861195
- [Background] Yamaguchi K, Martin CH, Boden SD, Labropoulos PA. Operative treatment of syndesmotic disruptions without use of a syndesmotic screw: a prospective clinical study. Foot Ankle Int. 1994 Aug;15(8):407-14. doi: 10.1177/107110079401500801. PMID 7981810
- [Background] Ramsey PL, Hamilton W. Changes in tibiotalar area of contact caused by lateral talar shift. J Bone Joint Surg Am. 1976 Apr;58(3):356-7. PMID 1262367
- [Background] Parfenchuck TA, Frix JM, Bertrand SL, Corpe RS. Clinical use of a syndesmosis screw in stage IV pronation-external rotation ankle fractures. Orthop Rev. 1994 Aug;Suppl:23-8. PMID 7970880
- [Background] Bauer M, Jonsson K, Nilsson B. Thirty-year follow-up of ankle fractures. Acta Orthop Scand. 1985 Apr;56(2):103-6. doi: 10.3109/17453678508994329. PMID 3925709
- [Background] Gardner MJ, Demetrakopoulos D, Briggs SM, Helfet DL, Lorich DG. Malreduction of the tibiofibular syndesmosis in ankle fractures. Foot Ankle Int. 2006 Oct;27(10):788-92. doi: 10.1177/107110070602701005. PMID 17054878
- [Background] Phillips WA, Schwartz HS, Keller CS, Woodward HR, Rudd WS, Spiegel PG, Laros GS. A prospective, randomized study of the management of severe ankle fractures. J Bone Joint Surg Am. 1985 Jan;67(1):67-78. PMID 3881447
- [Background] Coetzee JC, Ebeling P. Treatment of syndesmosis disruptions with TightRope Fixation. Tech Foot Ankle Surg. 7(3):196-202, 2008.
- [Background] Forsythe K, Freedman KB, Stover MD, Patwardhan AG. Comparison of a novel FiberWire-button construct versus metallic screw fixation in a syndesmotic injury model. Foot Ankle Int. 2008 Jan;29(1):49-54. doi: 10.3113/FAI.2008.0049. PMID 18275736
- [Background] Soin SP, Knight TA, Dinah AF, Mears SC, Swierstra BA, Belkoff SM. Suture-button versus screw fixation in a syndesmosis rupture model: a biomechanical comparison. Foot Ankle Int. 2009 Apr;30(4):346-52. doi: 10.3113/FAI.2009.0346. PMID 19356360
- [Background] Gardner MJ, Brodsky A, Briggs SM, Nielson JH, Lorich DG. Fixation of posterior malleolar fractures provides greater syndesmotic stability. Clin Orthop Relat Res. 2006 Jun;447:165-71. doi: 10.1097/01.blo.0000203489.21206.a9. PMID 16467626
- [Background] Klitzman R, Zhao H, Zhang LQ, Strohmeyer G, Vora A. Suture-button versus screw fixation of the syndesmosis: a biomechanical analysis. Foot Ankle Int. 2010 Jan;31(1):69-75. doi: 10.3113/FAI.2010.0069. PMID 20067726
- [Background] Miller RS, Weinhold PS, Dahners LE. Comparison of tricortical screw fixation versus a modified suture construct for fixation of ankle syndesmosis injury: a biomechanical study. J Orthop Trauma. 1999 Jan;13(1):39-42. doi: 10.1097/00005131-199901000-00009. PMID 9892124
- [Background] Ogilvie-Harris DJ, Reed SC, Hedman TP. Disruption of the ankle syndesmosis: biomechanical study of the ligamentous restraints. Arthroscopy. 1994 Oct;10(5):558-60. doi: 10.1016/s0749-8063(05)80014-3. PMID 7999167
- [Background] Miller AN, Carroll EA, Parker RJ, Boraiah S, Helfet DL, Lorich DG. Direct visualization for syndesmotic stabilization of ankle fractures. Foot Ankle Int. 2009 May;30(5):419-26. doi: 10.3113/FAI-2009-0419. PMID 19439142
- [Background] Pelton K, Thordarson DB, Barnwell J. Open versus closed treatment of the fibula in Maissoneuve injuries. Foot Ankle Int. 2010 Jul;31(7):604-8. doi: 10.3113/FAI.2010.0604. PMID 20663427
- [Background] Miller AN, Carroll EA, Parker RJ, Helfet DL, Lorich DG. Posterior malleolar stabilization of syndesmotic injuries is equivalent to screw fixation. Clin Orthop Relat Res. 2010 Apr;468(4):1129-35. doi: 10.1007/s11999-009-1111-4. Epub 2009 Oct 2. PMID 19798540